CLINICAL TRIAL: NCT01359800
Title: A Multicentre, Observational, Cross-sectional Study to Assess the Seroprevalence of Anti-Tat Antibodies in HIV-infected Patients in Selected Areas of Gauteng and Eastern Cape
Brief Title: Study to Assess the Seroprevalence of Anti-Tat Antibodies in HIV-infected Patients
Acronym: ISS OBS T-004
Status: Completed | Type: Observational
Sponsor: Barbara Ensoli, MD (Other)
Collaborators: Italian Ministry of Foreign Affairs - Dir. Gen. for Cooperation and Development (Unknown)
Responsible Party: Sponsor-Investigator, Barbara Ensoli, MD, PhD, Istituto Superiore di Sanità
Organization: Istituto Superiore di Sanità (Other)
Other Study IDs: ISS OBS T-004
Record Dates: First submitted 2011-05-17; First posted 2011-05-25 (Estimated); Last update posted 2016-03-04 (Estimated); Status verified 2016-03

CONDITIONS: HIV Infection
Keywords: HIV; HAART
MeSH Terms: conditions — HIV Infections

STUDY DESIGN:
Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Whole blood, cervical samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Treatment-naive HIV+ subjects
- HAART-treated HIV+ subjects

SUMMARY:
Tat is a key HIV regulatory protein produced very early after infection, prior to virus integration, and necessary for viral gene expression, cell-to-cell virus transmission and disease progression. Previous studies in natural HIV infection, indicated that the presence of a Tat-specific immune response correlates with a lower incidence and reduced risk of progression to AIDS as compared to anti-Tat negative individuals suggesting that an immune response to Tat may exert a protective role and control the progression to AIDS in vivo.

On the basis of the above mentioned consideration, the present study was directed at investigating the seroprevalence of anti-Tat antibodies in HIV-infected South African patients.

DETAILED DESCRIPTION:
This is an observational, cross-sectional study aimed at assessing the frequency, magnitude and quality of the anti-Tat antibody response in both antiretroviral (ARV)-treated and treatment-naïve HIV-infected South African adults, and at exploring the correlation between the presence of anti-Tat antibody response and the immunological status of participants as well as with the presence of co-infections such as HBV, syphilis and HPV (the latter only for female participants).

The study has involved 531 participants and provided important information for the planning, design and conduction of future therapeutic clinical trials with the Tat-based HIV vaccine in South African individuals.

This study is conducted in the frame of the Government-to-Government cooperation program N. AID 8421, funded by the Italian Ministry of Foreign Affairs-Directorate General for Development Cooperation (MAE-DGCS) and jointly implemented by the Italian Istituto Superiore di Sanita' (ISS) and the South African Department of Health in collaboration with the South African AIDS Vaccine Initiative of the Medical Research Council (MRC-SAAVI)

ELIGIBILITY:
Inclusion Criteria:

* HIV-infected individuals Aged 18-45 years Participants enrolled into the ARV-treated group must have been on treatment for not less than 3 months.

Exclusion Criteria:

* Unwillingness to consent to study inclusion

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: HIV positive, ARV-treated and treatment-naïve participants.
Sampling Method: Non-Probability Sample
Enrollment: 531 (Actual)
Dates: Start 2010-10; Primary Completion 2013-02 (Actual); Study Completion 2013-07 (Actual)

PRIMARY OUTCOMES:
Anti-Tat Antibody Responses | Up to 14 months
  Assessment of serum anti-Tat antibodies. Anti-Tat humoral immune response will include the determination of serum IgM, IgG and IgA antibodies against both clade B- and C-derived Tat proteins and titration of IgM, IgG and IgA anti-Tat antibodies.

SECONDARY OUTCOMES:
Virological status of anti-Tat positive and negative participants | Up to 14 months
  HIV viral load and clinical status on anti-Tat+ versus anti-Tat- participants. The effect of ARV treatment non-compliance on viral load in anti-Tat+ versus anti-Tat- participants has been evaluated within the ARV-treated study group on the basis of the relevant available information.
  Hepatitis B, Syphilis, HPV co-infections Assessment.
Immunological status of anti-Tat positive and negative participants | Up to 14 months
  Assessment of CD4 T cell counts. Exploratory immunological assays may be performed on available residual samples for a more in-depth characterisation of the immune response.
Immune activation status of anti-Tat positive and negative participants | Up to 14 months
  Assessment of Immune-activation markers on CD4+ and CD8+ T cells (CD25+, CD38+ and HLA-DR+).

CONTACTS AND LOCATIONS:
Overall Officials: Barbara BE Ensoli, MD PhD, Study Director — Istituto Superiore di Sanità
Locations (2):
- South Africa (2):
  - Walter Sisulu University HIV Vaccine Research Unit, Mthatha, Eastern Cape
  - Mecru Clinical Research Unit (MeCRU), Medunsa, Gauteng

REFERENCES:
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Tripiciano A, Longo O, Bellino S, Francavilla V, Paniccia G, Arancio A, Scoglio A, Collacchi B, Ruiz Alvarez MJ, Tambussi G, Tassan Din C, Palamara G, Latini A, Antinori A, D'Offizi G, Giuliani M, Giulianelli M, Carta M, Monini P, Magnani M, Garaci E. The preventive phase I trial with the HIV-1 Tat-based vaccine. Vaccine. 2009 Dec 11;28(2):371-8. doi: 10.1016/j.vaccine.2009.10.038. Epub 2009 Oct 29. PMID 19879233
- [Background] Longo O, Tripiciano A, Fiorelli V, Bellino S, Scoglio A, Collacchi B, Alvarez MJ, Francavilla V, Arancio A, Paniccia G, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Phase I therapeutic trial of the HIV-1 Tat protein and long term follow-up. Vaccine. 2009 May 26;27(25-26):3306-12. doi: 10.1016/j.vaccine.2009.01.090. Epub 2009 Feb 7. PMID 19208456
- [Background] Ensoli B, Bellino S, Tripiciano A, Longo O, Francavilla V, Marcotullio S, Cafaro A, Picconi O, Paniccia G, Scoglio A, Arancio A, Ariola C, Ruiz Alvarez MJ, Campagna M, Scaramuzzi D, Iori C, Esposito R, Mussini C, Ghinelli F, Sighinolfi L, Palamara G, Latini A, Angarano G, Ladisa N, Soscia F, Mercurio VS, Lazzarin A, Tambussi G, Visintini R, Mazzotta F, Di Pietro M, Galli M, Rusconi S, Carosi G, Torti C, Di Perri G, Bonora S, Ensoli F, Garaci E. Therapeutic immunization with HIV-1 Tat reduces immune activation and loss of regulatory T-cells and improves immune function in subjects on HAART. PLoS One. 2010 Nov 11;5(11):e13540. doi: 10.1371/journal.pone.0013540. PMID 21085635
- [Background] Bellino S, Francavilla V, Longo O, Tripiciano A, Paniccia G, Arancio A, Fiorelli V, Scoglio A, Collacchi B, Campagna M, Lazzarin A, Tambussi G, Din CT, Visintini R, Narciso P, Antinori A, D'Offizi G, Giulianelli M, Carta M, Di Carlo A, Palamara G, Giuliani M, Laguardia ME, Monini P, Magnani M, Ensoli F, Ensoli B. Parallel conduction of the phase I preventive and therapeutic trials based on the Tat vaccine candidate. Rev Recent Clin Trials. 2009 Sep;4(3):195-204. doi: 10.2174/157488709789957529. PMID 20028332
- [Background] Ensoli B, Fiorelli V, Ensoli F, Lazzarin A, Visintini R, Narciso P, Di Carlo A, Monini P, Magnani M, Garaci E. The therapeutic phase I trial of the recombinant native HIV-1 Tat protein. AIDS. 2008 Oct 18;22(16):2207-9. doi: 10.1097/QAD.0b013e32831392d4. PMID 18832884
- [Background] Ensoli B, Fiorelli V, Ensoli F, Cafaro A, Titti F, Butto S, Monini P, Magnani M, Caputo A, Garaci E. Candidate HIV-1 Tat vaccine development: from basic science to clinical trials. AIDS. 2006 Nov 28;20(18):2245-61. doi: 10.1097/QAD.0b013e3280112cd1. No abstract available. PMID 17117011
- [Background] Butto S, Fiorelli V, Tripiciano A, Ruiz-Alvarez MJ, Scoglio A, Ensoli F, Ciccozzi M, Collacchi B, Sabbatucci M, Cafaro A, Guzman CA, Borsetti A, Caputo A, Vardas E, Colvin M, Lukwiya M, Rezza G, Ensoli B; Tat Multicentric Study Group. Sequence conservation and antibody cross-recognition of clade B human immunodeficiency virus (HIV) type 1 Tat protein in HIV-1-infected Italians, Ugandans, and South Africans. J Infect Dis. 2003 Oct 15;188(8):1171-80. doi: 10.1086/378412. Epub 2003 Sep 30. PMID 14551888
- [Background] Rezza G, Fiorelli V, Dorrucci M, Ciccozzi M, Tripiciano A, Scoglio A, Collacchi B, Ruiz-Alvarez M, Giannetto C, Caputo A, Tomasoni L, Castelli F, Sciandra M, Sinicco A, Ensoli F, Butto S, Ensoli B. The presence of anti-Tat antibodies is predictive of long-term nonprogression to AIDS or severe immunodeficiency: findings in a cohort of HIV-1 seroconverters. J Infect Dis. 2005 Apr 15;191(8):1321-4. doi: 10.1086/428909. Epub 2005 Mar 14. PMID 15776379
- [Background] Bellino S, Tripiciano A, Picconi O, Francavilla V, Longo O, Sgadari C, Paniccia G, Arancio A, Angarano G, Ladisa N, Lazzarin A, Tambussi G, Nozza S, Torti C, Foca E, Palamara G, Latini A, Sighinolfi L, Mazzotta F, Di Pietro M, Di Perri G, Bonora S, Mercurio VS, Mussini C, Gori A, Galli M, Monini P, Cafaro A, Ensoli F, Ensoli B. The presence of anti-Tat antibodies in HIV-infected individuals is associated with containment of CD4+ T-cell decay and viral load, and with delay of disease progression: results of a 3-year cohort study. Retrovirology. 2014 Jun 24;11:49. doi: 10.1186/1742-4690-11-49. PMID 24961156
- [Background] Ensoli B, Cafaro A, Monini P, Marcotullio S, Ensoli F. Challenges in HIV Vaccine Research for Treatment and Prevention. Front Immunol. 2014 Sep 8;5:417. doi: 10.3389/fimmu.2014.00417. eCollection 2014. PMID 25250026
- [Background] Ensoli F, Cafaro A, Casabianca A, Tripiciano A, Bellino S, Longo O, Francavilla V, Picconi O, Sgadari C, Moretti S, Cossut MR, Arancio A, Orlandi C, Sernicola L, Maggiorella MT, Paniccia G, Mussini C, Lazzarin A, Sighinolfi L, Palamara G, Gori A, Angarano G, Di Pietro M, Galli M, Mercurio VS, Castelli F, Di Perri G, Monini P, Magnani M, Garaci E, Ensoli B. HIV-1 Tat immunization restores immune homeostasis and attacks the HAART-resistant blood HIV DNA: results of a randomized phase II exploratory clinical trial. Retrovirology. 2015 Apr 29;12:33. doi: 10.1186/s12977-015-0151-y. PMID 25924841
- [Background] Cafaro A, Tripiciano A, Sgadari C, Bellino S, Picconi O, Longo O, Francavilla V, Butto S, Titti F, Monini P, Ensoli F, Ensoli B. Development of a novel AIDS vaccine: the HIV-1 transactivator of transcription protein vaccine. Expert Opin Biol Ther. 2015;15 Suppl 1:S13-29. doi: 10.1517/14712598.2015.1021328. Epub 2015 Jun 22. PMID 26096836
- See also: Related Info — http://www.hiv1tat-vaccines.info